CLINICAL TRIAL: NCT01075945
Title: Dihydroartemisinin- Piperaquine Versus Artemether- Lumefantrine in the Treatment Uncomplicated Plasmodium Falciparum Malaria in Sudan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Khartoum (Other)
Collaborators: Southeast University, China (Other)
Responsible Party: Prof., Univeristy of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP v AL01; DP v AL01aasudan (Other: Holley); wadadam
Record Dates: First submitted 2010-02-18; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Malaria
Keywords: antimalarials; ACTs; Piperaquine; uncomplicated
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dihydroartemisinin- piperaquine (Experimental): orally tablets
  Interventions: Drug: Dihydroartemisinin- piperaquine; Drug: artemether- lumefantrine
- artemether- lumefantrine (Active Comparator): oral tablets
  Interventions: Drug: artemether- lumefantrine

INTERVENTIONS:
Drug: Dihydroartemisinin- piperaquine — three tablets per day
  Other Names: Hoy-Cotec
  Arms: Dihydroartemisinin- piperaquine
Drug: artemether- lumefantrine — twenty tablet in eight doses
  Other Names: Coartem

SUMMARY:
Dihydroartemisinin- Piperaquine is not inferior to artemether-lumefantrine

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated malaria

Exclusion Criteria:

* Severe cases
* Pregnancy

Ages: 5 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
comparing the cure rate between the two drugs | 3 months
  PCR cure rate Parasite clearance time Fever clearance time

CONTACTS AND LOCATIONS:
Locations (1):
- Sinnar, Cinnar, Blue Nile, Sudan

REFERENCES:
- [Background] Adam I, Elmardi KA, Malik EM. Predictors of antimalarial treatment failure in an area of unstable malaria transmission in eastern Sudan. Trans R Soc Trop Med Hyg. 2009 Jan;103(1):21-4. doi: 10.1016/j.trstmh.2008.07.005. Epub 2008 Aug 20. PMID 18718621